CLINICAL TRIAL: NCT02312466
Title: Swiss National Iodine Survey 2015; A Cross-sectional Study to Assess Iodine Status in School Children, Women of Reproductive Age and Pregnant Women
Brief Title: Swiss National Iodine Survey 2015
Acronym: SIS
Status: Completed | Type: Observational
Sponsor: Isabelle Herter-Aeberli (Other)
Collaborators: Federal Food Safety and Veterinary Office (Switzerland) (Unknown)
Responsible Party: Sponsor-Investigator, Isabelle Herter-Aeberli, PhD, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Other Study IDs: SIS 2015
Record Dates: First submitted 2014-12-03; First posted 2014-12-09 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- School aged children
- Pregnant women
- Women of reproductive age

SUMMARY:
The aim of this study is to monitor iodine nutrition in Switzerland in order to inform the authorities regarding iodine content in iodized salt. As a proxy for the entire population the investigators will study school aged children, pregnant women and women of reproduction age.

DETAILED DESCRIPTION:
In a national sample of school aged children (n=990), pregnant women (n=700) and women of reproductive age (n=700) urinary iodine will be determined in order to assess iodine nutrition in Switzerland. In addition, in both groups of women a blood sample will be taken for the determination of thyroid hormones, iron- and folate status. Questionnaires will be used for the determination of dietary iodine and salt intake as well as sociodemographic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Living in Switzerland for at least 1 year
* For pregnant women: singleton pregnancy

Exclusion Criteria:

* Major known medical illness: thyroid dysfunction, gastrointestinal or metabolic disorders and taking chronic medications
* For women of reproductive age: pregnancy, breastfeeding
* Use of X-ray or CT contrast agent or iodine containing medication within the past year

Ages: 6 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: school aged children, 6-12 years pregnant women, 18-44 years women of reproductive age, 18-44 years
Sampling Method: Probability Sample
Enrollment: 1430 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Median urinary iodine concentration in school aged children, pregnant women and women of reproductive age | Baseline
  analysis of urine samples

SECONDARY OUTCOMES:
Population mean thyroglobulin | Baseline
  Analysis of venous blood samples. Assessed only in women
Population mean thyroid stimulating hormone | Baseline
  Analysis of venous blood samples. Assessed only in women
Population mean thyroxine | Baseline
  Analysis of venous blood samples. Assessed only in women
Median urinary sodium concentration | Baseline
Median urinary creatinin concentration | Baseline

OTHER OUTCOMES:
Mean height of school aged children and women of reproductive age | Baseline
Mean weight of school aged children and women of reproductive age | Baseline
Median urinary fluoride | Baseline
  Analyzed in urine samples from school aged children only.
Population mean folate status | Baseline
  Analysis of red blood cell folate and plasma folate in venous blood samples.
Populations mean iron status | Baseline
  Serum analysis: ferritin, transferrin receptor; in women of reproductive age and pregnant women.
Individual inflammatory state | Baseline
  Serum analysis of CRP and AGP, analyzed only in women
Intake of iodine in micro grams per day | Baseline
  iodine intake assessed by food frequency questionnaire, only in women
% of households with adequate iodine coverage | Baseline
  Salt samples only collected from children (subgroup)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Laboratory, ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Andersson M, Hunziker S, Fingerhut R, Zimmermann MB, Herter-Aeberli I. Effectiveness of increased salt iodine concentration on iodine status: trend analysis of cross-sectional national studies in Switzerland. Eur J Nutr. 2020 Mar;59(2):581-593. doi: 10.1007/s00394-019-01927-4. Epub 2019 Mar 1. PMID 30843107